CLINICAL TRIAL: NCT03882593
Title: Blood Cell Adhesion to Arterial Filters During Cardic Surgery - Observational Clinical Study: Scanning Electron Microscopy and Cell Gene Expression Analysis
Brief Title: Blood Cell Adhesion to Arterial Filters During Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Instituto do Coracao (Other Government)
Responsible Party: Principal Investigator, Filomena R B G Galas, Associate Professor of Anesthesiology at University São Paulo Medical School, Instituto do Coracao
Other Study IDs: 4279.15.106
Record Dates: First submitted 2018-08-30; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Blood Coagulation Disorders; C.Surgical Procedure; Cardiac
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Analysis of arterial filters during CPB: This is a clinical and observational study to investigate of blood cells addesion to surfaces of arterial filters during CPB and the impact in coagulations laboratory exams
  Interventions: Procedure: Analysis of arterial filters after CPB

INTERVENTIONS:
Procedure: Analysis of arterial filters after CPB — At the end of surgery, the arterial filter is withdrawn from cardiopulmonary bypass circuit to be prepared and analysed by SEM.

SUMMARY:
Cardiopulmonary bypass (CPB) is a unique clinical scenario that results in widespread activation of the hemostatic system. Conventional CPB interferes with normal hemostasis by diluting hemostatic cells and proteins, through reinfusion of shed blood, and through activation on the bypass circuit surface of multiple systems including platelets, the kallikrein-kinin system, and fibrinolysis . Besides, deleterious effects of cardiopulmonary bypass (CPB) are partly sequelae of blood-foreign surface reactions. The arterial filter is the part of the CPB circuit where blood cells are exposed to high mechanical stress and where cellular aggregates may fasten in large quantitiesiec.

DETAILED DESCRIPTION:
This is a clinical and observational study. It is being performed in the surgical center and intensive care unit of the Heart Institute (InCor) from Faculty of Medicine, University of São Paulo (FMUSP), on patients undergoing cardiac surgery, who satisfy inclusion and exclusion criteria. In the preanesthetic visit, patient assessment of the criteria described in study methodology is verfied. During the surgery, a blood sample is taken to analyze hemostatic function in the begin of cardiopulmonary bypass, before arterial filter (pre-filter) and in the end of cardiopulmonary bypass, after arterial filter (post-filter). Other routine laboratory exams is being colected until first postoperative day, on the eletronic medical records. At the end of surgery, the arterial filter is withdrawn from cardiopulmonary bypass circuit to be prepared and analysed by SEM. Ten arterial filter samples from pre-determined sites and sizes are sent to the clinical laboratory for evaluation of platelet and leukocyte gene expression in arterial filter. Patients will be followed until hospital discharge or 28 days after surgery, regarding allogeneic transfusion needs, reoperation and thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgeries with extracorporeal circulation in patients older than 18 years
* Written and signed informed consent
* Preanesthetic assessment and preoperatory exams in accordance with study methodology

Exclusion Criteria:

* Active infection;
* Previously coagulopathy;
* Antiplatelet therapy use until 10 days before surgery (except acetylsalicylic acid and enoxaparin that may be used in prophylactic doses until 24h before surgery);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery with cardiopulmonary bypass (CPB)
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-05 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Types and characteristics of materials entrapped in the arterial line filter of cardiopulmonary bypass | At the beginning and end of cardiopulmonary bypass
  Analysis of the arterial filter from cardiopulmonay bypass circuit by scanning electron microscopy (SEM)
Platelet and leukocyte gene expression analysis of arterial line filters of cardiopulmonary bypass | At the beginning and end of cardiopulmonary bypass
  Arterial filter samples from predetermined sites and sizes will be analyzed for evaluation of platelet and leukocyte gene expression in arterial filter.

SECONDARY OUTCOMES:
Correlation between blood adhesion cells in arterial filter and coagulation tests | At the beginning and end of cardiopulmonary bypass
Comparison of standard coagulation test | At the beginning and end of cardiopulmonary bypass, Immediate postoperative; 24 hours and 48 hours after surgery
  Analysis of coagulation profile will be assessed fibrinogen dosage (mg/dL), D-dimers (ng/mL), hemoglobin(g/dL), hematocrit (%), platelets count (mm³), prothrombin time (s), activated thromboplastin time (s), international normalized ratio.
Comparison of free oscillation rheometry profile | At the beginning and end of cardiopulmonary bypass
  Analysis of HEPSCREEN (Reorox) COT1(s),COT2(s), Slope (Pa/min), GMAX (Pa), EAT (Pa), CLOT SR(%)

CONTACTS AND LOCATIONS:
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Reynolds PS, Middleton P, McCarthy H, Spiess BD. A Comparison of a New Ultrasound-Based Whole Blood Viscoelastic Test (SEER Sonorheometry) Versus Thromboelastography in Cardiac Surgery. Anesth Analg. 2016 Dec;123(6):1400-1407. doi: 10.1213/ANE.0000000000001362. PMID 27159065
- [Background] Borowiec JW, Bylock A, van der Linden J, Thelin S. Heparin coating reduces blood cell adhesion to arterial filters during coronary bypass: a clinical study. Ann Thorac Surg. 1993 Jun;55(6):1540-5. doi: 10.1016/0003-4975(93)91106-w. PMID 8512409
- [Background] Galas FR, de Almeida JP, Fukushima JT, Vincent JL, Osawa EA, Zeferino S, Camara L, Guimaraes VA, Jatene MB, Hajjar LA. Hemostatic effects of fibrinogen concentrate compared with cryoprecipitate in children after cardiac surgery: a randomized pilot trial. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1647-55. doi: 10.1016/j.jtcvs.2014.04.029. Epub 2014 Apr 18. PMID 24951020